CLINICAL TRIAL: NCT06033872
Title: Effectiveness of Diabetes Education and Medication Adjustment With Telemonitoring Intervention in Reducing Diabetes Complications During Ramadan Fasting - a Randomized Control Trial
Brief Title: Effectiveness of Education, Medication Adjustment and Telemonitoring in Reducing Diabetes Complications During Ramadan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sengkang General Hospital (Other)
Collaborators: SingHealth Polyclinics (Other); Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/2888
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus; Fasting; Diabetes Complications
MeSH Terms: conditions — Diabetes Mellitus; Fasting; Diabetes Complications

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Focused education, medication adjustment and telemonitoring
  Interventions: Combination Product: Focused education, medication adjustment and telemonitoring
- Control (No Intervention): Standard care

INTERVENTIONS:
Combination Product: Focused education, medication adjustment and telemonitoring — 1. Focused diabetes education session for Ramadan fasting
     Participants will be taught to record
     1. Meal plans
     2. Physical activities
     3. Blood glucose monitoring, and
     4. Monitoring for diabetes complications. Then perform a trial fasting day prior to Ramadan when control is not optimal or medication with risk of hypoglycemia.
  2. Medication adjustment for Ramadan fasting Participants will be provided regimen modified for Ramadan fasting.
  3. Telemonitoring
  Participants will be taught to perform blood glucose monitoring 4 times daily using a glucometer and upload recordings of glucose levels onto the data software.
  Arms: Intervention

SUMMARY:
Introduction Diabetes is a global emergency with detrimental clinical and financial consequences. Poorly managed diabetes leads to a myriad of serious complications, especially cardiovascular and infectious complications, with consequent increased cost and mortality rate. For Muslims in particular, the annual fasting month of Ramadan is one such period when diabetes control is essential. Adequate adjustments in diabetes management need to be made in line with the allowed meal times to avoid the risk of diabetes complications during Ramadan.

Objective Investigators aim to investigate the effectiveness of focused diabetes education and medication adjustment with telemonitoring to reduce diabetes complications during Ramadan fasting as well as to assess the cost-effectiveness of this intervention for Muslims with diabetes in Singapore.

Methodology In a parallel group randomized controlled trial, investigators aim to recruit 100 adults with diabetes who are able to fast at least 15 days in Ramadan. Participants will be randomized to the intervention group comprising of focused diabetes education, medication adjustment and telemonitoring, and control group receiving standard care. Participants will be followed up during Ramadan. The primary outcome is the incidence of hypoglycemia in Ramadan. The secondary outcomes are (i) incidence of other diabetes complications in Ramadan episodes including hyperglycemia, episodes of acute infections, attendances in clinic and emergency department and that of hospital admission, and (ii) cost-effectiveness of the intervention.

Clinical Significance The study enables investigators to evaluate focused pre-Ramadan diabetes education and medication adjustment with tele-monitoring as a means to reduce the markedly increased risk of diabetes complications for a large population during the fasting month, with potential for increased cost-effectiveness through reducing unscheduled attendances at clinic and hospital.

ELIGIBILITY:
Inclusion Criteria:

-

Participants must meet all of the inclusion criteria to participate in this study:

1. Adults aged at least 21 years old,
2. Able to fast at least 15 days in Ramadan based on experience of fasting in previous year's Ramadan,
3. Known physician-diagnosed diabetes mellitus (DM) based on the following criteria before starting treatment

   a. Symptoms of polyuria, polydipsia and unexplained weight loss with i. fasting glucose ≥ 7.0mmol/l or ii. random plasma glucose ≥ 11.1 mmol/l or iii. 2-hour post 75g oral glucose challenge test plasma glucose ≥ 11.1 mmol/l b. Absence of symptoms of polyuria, polydipsia and unexplained weight loss with the following tests done twice showing the values i. fasting glucose ≥ 7.0mmol/l or ii. random plasma glucose ≥ 11.1 mmol/l or iii. 2-hour post 75g oral glucose challenge test plasma glucose ≥ 11.1 mmol/l
4. Performed laboratory tests as per standard care : serum glycated hemoglobin A1c (HbA1c) level, blood Low Density Lipoprotein-Cholesterol, blood triglyceride level, blood High Density Lipoprotein-Cholesterol, blood Total Cholesterol and serum creatinine
5. Most recent HbA1c level was >7.0% (>53mmol/mol)
6. Ability to give informed consent,
7. Ability to perform weekly recordings in the diary,
8. Able to use and owns a mobile phone for recordings on mobile application
9. Should have had DM-related clinic visits or hospitalization in the past 10 months.

Exclusion Criteria:

-

Meeting any of the exclusion criteria at baseline will exclude participants from participation:

1. Severe diabetes complications including end-stage renal failure, severe hypoglycemia and hyperglycemic crises within the last 1 month negating ability to fast,
2. Pregnancy.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
a. To compare the first incidence rate of hypoglycemia or severe hypoglycemia between intervention and control groups in Ramadan | 30 day

SECONDARY OUTCOMES:
i. To compare the first incidence rate of hypoglycemia or severe hypoglycemia between intervention and control groups in Ramadan when compared to before and after Ramadan | 12 weeks
ii. To compare the first incidence rate of complications in Ramadan when compared to before and after 1. Hyperglycemia and crises 2. Acute infections, clinic and emergency department attendances and hospital admissions | 12 weeks
Health-related Quality-of-Life using European Quality of Life Five Dimensions (EQ-5D) - to provide a summary of index value of health and health change, cost-utility calculation. | 17 weeks
  Five dimensions are mobility, self-care, usual activities, pain or discomfort and anxiety or depression. Scored health as 0 to 100 where 0 is worst and 100 is best
Healthcare utilizations costs - Medical services, drugs and devices utilized, outpatient and inpatient visits, cost of intervention sessions, telemonitoring and equipment, indirect costs related to health care utilisation, and caregiver costs. | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sueziani B Zainudin, MBBS FRCPG, Principal Investigator — Sengkang General Hospital
Locations (1):
- Sengkang General Hospital, Singapore, Singapore